CLINICAL TRIAL: NCT02141035
Title: Acetyl-l-carnitine to Enhance Nerve Regeneration in Carpal Tunnel Syndrome; a Randomized Control Trial.
Brief Title: Acetyl-l-carnitine to Enhance Nerve Regeneration in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Ming Chan, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00045538; RES0021133 (Other Grant/Funding Number: University of Alberta Hospital Foundation)
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Carpal Tunnel Syndrome; Compression Neuropathy
Keywords: Acetyl-l-carnitine; Carpal tunnel syndrome; Motor unit number estimation; Compression neuropathy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Tomaculous neuropathy | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetyl-l-carnitine (Experimental): Acetyl-l-carnitine will be administered for 2 months duration at a dosage of 3000 mg/d starting at the time of decompression surgery.
  Interventions: Drug: Acetyl-l-carnitine
- Placebo (Placebo Comparator): Placebo will be given for 2 months starting at the time of decompression surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Acetyl-l-carnitine — Those randomized to the treatment arm will receive the medication at 1 g tid for 60 days
  Arms: Acetyl-l-carnitine
Drug: placebo — The control subjects will receive placebo tablets that are identical in appearance and taste to the active medication tid for 60 days
  Arms: Placebo

SUMMARY:
Study Hypothesis: Acetyl-l-carnitine increases nerve regeneration in patients with severe carpal tunnel syndrome.

Carpal tunnel syndrome (CTS) is common, affecting almost 3% of the general population. In severe cases, nerve regeneration and functional recovery are incomplete even with surgery. The goal of this pilot project is to test a potentially promising medication, acetyl-l-carnitine (ALCAR). We will use a randomized, double blinded, placebo controlled study design. Along with surgery, those in the treatment group will also receive ALCAR while the other half in the control group will be given placebo. To gauge the effects of ALCAR, we will compare motor and sensory nerve growth as well as functional outcomes. The data from this study will provide crucial information when designing a full scale clinical trial. If successful, this will represent an important first step in finding a novel treatment to improve functional outcomes in patients with severe CTS.

DETAILED DESCRIPTION:
Trial Conduct: This study will be conducted in compliance with the protocol approved by both the University of Alberta Health Research Ethics Board (HREB) and Health Canada. The study will be carried out according to Good Clinical Practice standards. No deviation from the protocol will occur once approved, unless the protocol has put patients at risk. If deviation needs to occur, both HREB and Health Canada will be notified. Written amendments will be submitted to both HREB and Health Canada for their approval.

Population Adult patients suffering from severe CTS would be a population of the interest. Severity of CTS is defined by clinical symptoms and electromyography (EMG) results. These patients will then be recruited for baseline studies, motor unit number estimation (MUNE). Motor unit number estimation is an EMG technique that quantifies the amount of motor units a muscle contains. In various forms of neuropathies, the MUNE decreases. For our study, patients will be included only if their MUNE is 2 standard deviations below normal. These patients will be identified from referrals to plastic surgery clinics or EMG clinics for management.Pre-study Screening and Baseline Evaluation The subject will have a complete physical exam including clinical labs and an ECG. Only those who have normal laboratory and ECG findings will be enrolled in the study.

Randomization Randomization - After enrollment, patients will be randomized to placebo or acetyl-l-carnitine. A statistician will be employed to develop a randomization sequence. Randomization will be kept on a computer under password encryption. The randomization sequence will only be broken if an adverse event occurs to a patient. At the end of the study the statistician will provide the research team with the randomization sequence codes.

Blinding - The study will be administered in a double-blind manner. The randomization sequence will be kept confidential and only accessible to authorized personnel. Pharmacy will distribute identical pills labelled in bottles with A or B. The research team will be unaware of which contains the study drug or placebo. This will be maintained until the final follow-up has occurred when the research team will be unblinded.

Duration The duration of the study is approximately 13 months for each patient. Screening and baseline evaluation will occur within 1 month preoperatively. The investigators will review and document the screening laboratory tests and ECG results. Acetyl-l-carnitine regimen will begin immediately following surgery. This will be continued for 2 months duration. The patient will then complete follow-up visits at 1, 2, 3, 6, and 12 month intervals. At some of those visits, safety monitoring will include periodic blood chemistries, vital signs and evaluation of overall clinical condition (details shown in table above). All clinically relevant changes occurring during the study will be examined and documented. In cases where laboratory abnormalities are detected, appropriate medical management and advice will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the University of Alberta Hospital referred for CTS. Inclusion criteria will include adult patients (over age 18) with at least one of the following symptoms:

  1. numbness and parenthesis in the median nerve distribution;
  2. Precipitation of those symptoms by repetitive motions that are relieved by rubbing and or shaking the hands;
  3. Nocturnal awakening by those sensory symptoms, or
  4. Weakness of thumb abduction and thenar atrophy.

Exclusion Criteria:

1. Motor unit loss in the median nerve less than 2 SD below the mean for the age as determined by nerve conduction studies.
2. The presence of other neurologic conditions
3. Previous carpal tunnel release surgery
4. Cognitive impairment that renders the patient unable to provide informed consent;
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in motor unit number estimates | Baseline, 3, 6, and 12 months
  An electromyography technique used to quantify the number of motor units in a motor nerve.

SECONDARY OUTCOMES:
Change in two point discrimination | Baseline, 3, 6, and 12 months
  Measurement of spatial determination
Change in pressure sensitivity using Semmes-Weinstein Monofilaments | Baseline, 3, 6, and 12 months
  Measurement of pressure sensitivity
Change in cold detection threshold | Baseline, 3, 6, and 12 months
Change in pain detection thresholds | Baseline, 3, 6, and 12 months
  Quantitative measurements of pain thresholds
Change in hand dexterity using the Purdue Pegboard | Baseline, 3, 6, and 12 months
  Measurement of hand dexterity
Change in disability scores using the Disability of Arm, Shoulder and Hand questionnaire | Baseline, 3, 6, and 12 months
  Validated questionnaire for functionality in carpal tunnel syndrome
Change in hand symptoms using the Levine questionnaire for carpal tunnel syndrome | Baseline, 3, 6, and 12 months
  Validated questionnaire for functionality in carpal tunnel syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chan, MB,ChB, Principal Investigator — Professor, University of Alberta
Locations (3):
- Canada (3):
  - Glenrose Hosptial, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

REFERENCES:
- [Background] Atroshi I, Gummesson C, Johnsson R, McCabe SJ, Ornstein E. Severe carpal tunnel syndrome potentially needing surgical treatment in a general population. J Hand Surg Am. 2003 Jul;28(4):639-44. doi: 10.1016/s0363-5023(03)00148-5. PMID 12877853
- [Background] Barhwal K, Hota SK, Prasad D, Singh SB, Ilavazhagan G. Hypoxia-induced deactivation of NGF-mediated ERK1/2 signaling in hippocampal cells: neuroprotection by acetyl-L-carnitine. J Neurosci Res. 2008 Sep;86(12):2705-21. doi: 10.1002/jnr.21722. PMID 18500755
- [Background] Bianchi G, Vitali G, Caraceni A, Ravaglia S, Capri G, Cundari S, Zanna C, Gianni L. Symptomatic and neurophysiological responses of paclitaxel- or cisplatin-induced neuropathy to oral acetyl-L-carnitine. Eur J Cancer. 2005 Aug;41(12):1746-50. doi: 10.1016/j.ejca.2005.04.028. PMID 16039110
- [Background] Bitar G, Alexandrides J, Missirian R, Sotereanos D, Nystrom A. Carpal tunnel release in the United States and Sweden: reimbursement patterns, cost for treatment, and return to work. Plast Reconstr Surg. 2002 Apr 15;109(5):1574-8; discussion 1579-80. doi: 10.1097/00006534-200204150-00013. PMID 11932599
- [Background] Boyd JG, Gordon T. Neurotrophic factors and their receptors in axonal regeneration and functional recovery after peripheral nerve injury. Mol Neurobiol. 2003 Jun;27(3):277-324. doi: 10.1385/MN:27:3:277. PMID 12845152
- [Background] Bunge RP. Expanding roles for the Schwann cell: ensheathment, myelination, trophism and regeneration. Curr Opin Neurobiol. 1993 Oct;3(5):805-9. doi: 10.1016/0959-4388(93)90157-t. PMID 8260833
- [Background] Chen YY, McDonald D, Cheng C, Magnowski B, Durand J, Zochodne DW. Axon and Schwann cell partnership during nerve regrowth. J Neuropathol Exp Neurol. 2005 Jul;64(7):613-22. doi: 10.1097/01.jnen.0000171650.94341.46. PMID 16042313
- [Background] Grandis DD. Tolerability and efficacy of L-acetylcarnitine in patients with peripheral neuropathies: a short-term, open multicentre study. Clin Drug Investig. 1998;15(2):73-9. doi: 10.2165/00044011-199815020-00001. PMID 18370471
- [Background] De Grandis D, Minardi C. Acetyl-L-carnitine (levacecarnine) in the treatment of diabetic neuropathy. A long-term, randomised, double-blind, placebo-controlled study. Drugs R D. 2002;3(4):223-31. doi: 10.2165/00126839-200203040-00001. PMID 12455197
- [Background] Dudek H, Datta SR, Franke TF, Birnbaum MJ, Yao R, Cooper GM, Segal RA, Kaplan DR, Greenberg ME. Regulation of neuronal survival by the serine-threonine protein kinase Akt. Science. 1997 Jan 31;275(5300):661-5. doi: 10.1126/science.275.5300.661. PMID 9005851
- [Background] Evans JD, Jacobs TF, Evans EW. Role of acetyl-L-carnitine in the treatment of diabetic peripheral neuropathy. Ann Pharmacother. 2008 Nov;42(11):1686-91. doi: 10.1345/aph.1L201. Epub 2008 Oct 21. PMID 18940920
- [Background] Fu SY, Gordon T. Contributing factors to poor functional recovery after delayed nerve repair: prolonged denervation. J Neurosci. 1995 May;15(5 Pt 2):3886-95. doi: 10.1523/JNEUROSCI.15-05-03886.1995. PMID 7751953
- [Background] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Background] Gutmann E, Guttmann L, Medawar PB, & Young JZ (1942). The rate of regeneration of nerve. J Exp Biol 19, 14-44.
- [Background] Hall SM. The biology of chronically denervated Schwann cells. Ann N Y Acad Sci. 1999 Sep 14;883:215-33. PMID 10586247
- [Background] McKay Hart A, Wiberg M, Terenghi G. Pharmacological enhancement of peripheral nerve regeneration in the rat by systemic acetyl-L-carnitine treatment. Neurosci Lett. 2002 Dec 16;334(3):181-5. doi: 10.1016/s0304-3940(02)00982-5. PMID 12453625
- [Background] Kaplan DR, Miller FD. Neurotrophin signal transduction in the nervous system. Curr Opin Neurobiol. 2000 Jun;10(3):381-91. doi: 10.1016/s0959-4388(00)00092-1. PMID 10851172
- [Background] Kotil K, Kirali M, Eras M, Bilge T, Uzun H. Neuroprotective effects of acetyl-L-carnithine in experimental chronic compression neuropathy. A prospective, randomized and placebo-control trials. Turk Neurosurg. 2007 Apr;17(2):67-77. PMID 17935020
- [Background] Mazzoni IE, Said FA, Aloyz R, Miller FD, Kaplan D. Ras regulates sympathetic neuron survival by suppressing the p53-mediated cell death pathway. J Neurosci. 1999 Nov 15;19(22):9716-27. doi: 10.1523/JNEUROSCI.19-22-09716.1999. PMID 10559381
- [Background] Sulaiman OA, Gordon T. Effects of short- and long-term Schwann cell denervation on peripheral nerve regeneration, myelination, and size. Glia. 2000 Dec;32(3):234-46. doi: 10.1002/1098-1136(200012)32:33.0.co;2-3. PMID 11102965
- [Background] SUNDERLAND S. Rate of regeneration in human peripheral nerves; analysis of the interval between injury and onset of recovery. Arch Neurol Psychiatry. 1947 Sep;58(3):251-95. doi: 10.1001/archneurpsyc.1947.02300320002001. No abstract available. PMID 20265595
- [Background] Wilson AD, Hart A, Brannstrom T, Wiberg M, Terenghi G. Primary sensory neuronal rescue with systemic acetyl-L-carnitine following peripheral axotomy. A dose-response analysis. Br J Plast Surg. 2003 Dec;56(8):732-9. doi: 10.1016/j.bjps.2003.08.005. PMID 14615246
- [Background] You S, Petrov T, Chung PH, Gordon T. The expression of the low affinity nerve growth factor receptor in long-term denervated Schwann cells. Glia. 1997 Jun;20(2):87-100. doi: 10.1002/(sici)1098-1136(199706)20:23.0.co;2-1. PMID 9179594
- [Background] Youle M, Osio M; ALCAR Study Group. A double-blind, parallel-group, placebo-controlled, multicentre study of acetyl L-carnitine in the symptomatic treatment of antiretroviral toxic neuropathy in patients with HIV-1 infection. HIV Med. 2007 May;8(4):241-50. doi: 10.1111/j.1468-1293.2007.00467.x. PMID 17461852
- [Result] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Derived] Curran MW, Olson J, Morhart M, Sample D, Chan KM. Acetyl-L-carnitine (ALCAR) to enhance nerve regeneration in carpal tunnel syndrome: study protocol for a randomized, placebo-controlled trial. Trials. 2016 Apr 14;17:200. doi: 10.1186/s13063-016-1324-2. PMID 27079660